CLINICAL TRIAL: NCT03223974
Title: Clinical Trial on Safety and Efficacy of Drug-coated Balloon in Treatment of Coronary Bifurcation Lesions
Acronym: BJDCB-BIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xue Yu, Project manager, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJYY121-2016003
Record Dates: First submitted 2017-07-15; First posted 2017-07-21 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Coronary Disease
Keywords: Angioplasty; drug-coated balloon; bifurcation
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paclitaxel DCB for MB and/or SB (Experimental): Balloon/vessel diameter ratio 0.8-1.0, 8-10 ATM(atmosphere), lasting for >30 seconds
  Interventions: Device: Paclitaxel DCB
- DES in MB (Active Comparator): with regular techniques
  Interventions: Device: DES

INTERVENTIONS:
Device: Paclitaxel DCB — Balloon/vessel diameter ratio 0.8-1.0, 8-10 ATM, lasting for >30 seconds. If quantitative coronary angiography determines residual stenosis ≤ 30% , it is considered to be a successful operation.
  Arms: Paclitaxel DCB for MB and/or SB
Device: DES — MB should be sufficiently predilated to facilitate the positioning of the stent and the stent residual stenosis should be ≤10% to be a successful operation.
  Arms: DES in MB

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of paclitaxel-coated balloon in treatment of coronary bifurcation lesions. This is a feasible study to demonstrate the noninferiority of paclitaxel Drug-coated balloon(DCB) only strategy for bifurcation lesions when compared with traditional single drug eluting stent(DES) strategy, so as to simplify the procedure for treatment of coronary bifurcation lesions and extending the clinical indications of paclitaxel DCB in China.

DETAILED DESCRIPTION:
Paclitaxel DCB is designed to release anti-proliferative agents to the whole lesion rapidly and homogenously to inhibit excessive neointima proliferation and is associated with rapid healing of endothelium. As a result, DCB therapy reduces the risk of coronary thrombosis. Since only 1 to 3 months duration of dual anti-platelet therapy is required, the bleeding risk associated with prolonged dual anti-platelet therapy (DAPT) is reduced by DCB. Furthermore, there is no permanent residue of foreign bodies in the blood vessels after DCB procedure and this advantage completely eliminates adverse events associated with allergic reactions to metal, polymer and stent fracture. For side branch(SB) with a relatively small lumen in bifurcation lesions, DCB may neglect the lumen loss due to stent scaffolds and cause much less late lumen loss (LLL) than stent therapy does. For main branch(MB), no jailed SBs by the stent and the rate of SB stenosis or even occlusion will be greatly reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria：

  * Patients with stable angina, unstable angina, old myocardial infarction or evidence of asymptomatic myocardial ischemia and consent to receive coronary intervention therapy;
  * Aged between 18 and 80 years;
  * Consent to receive angiographic follow up at 9 months and clinical follow up at 30 days, 6, 9, 12 and 24 months.
* Lesion-related criteria：

  * Target lesions of Medina (0,1,1), (1,0,1) or (1,1,1) primary coronary bifurcation lesions without previous intervention therapy;
  * MB reference vessel diameter between 2.5 mm and 3.5 mm and length ≤30mm; SB reference vessel diameter between 2.0 mm and 3.0 mm and length ≤22 mm;
  * Pre-operative vessel diameter stenosis must ≥70% or ≥50% associated with local ischemia;
  * After lesion predilation, no dissection is seen, or type A/B dissection can be seen, residual stenosis ≤30% and TIMI(thrombolysis in myocardial infarction) grade 3 flow;
  * The distance between other lesions requiring intervention therapy and the target lesion must >10mm ;
  * Only one drug-eluting balloon or drug-eluting stent is used in treatment of MB and SB lesions.

Exclusion Criteria:

* Patient-related criteria：

  * Myocardial infarction in the previous week;
  * Severe congestive heart failure[LVEF <30% or NYHA( New York Heart Association) III/IV)]
  * Severe valvular heart disease;
  * Pregnant or breastfeeding women;
  * Life expectancy no more than 1 year or factors causing difficulties in clinical follow up;
  * Bleeding predisposition, contraindications of anticoagulants or antiplatelet agents;
  * Intolerance to aspirin and/or clopidogrel;
  * Known intolerance or allergy to heparin, contrast agents, paclitaxel, iopromide, rapamycin, polylactic acid-glycolic acid copolymer, Co-Cr alloy or platinum-chromium alloy;
  * Leukopenia or thrombopenia;
  * A history of peptic ulcer or GI bleeding in the previously;
  * Stroke within 6 months prior to the operation;
  * A history of severe hepatic or renal failure.
* Lesion-related criteria ：

  * Extensive thrombosis in the target vessel;
  * Percutaneous coronary intervention of the graft vessel;
  * Chronic total occlusions (pre-operative TIMI grade 0 flow);
  * Left main branch lesions and /or three-vessel lesions requiring treatment;
  * Lesions that are not indications of PTCA(percutaneous transluminal coronary angiography) or other intervention therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
QCA(quantitative coronary analysis) of efficacy of DCB | Follow-up coronary angiography at 9 months after the procedure
  late lumen loss, minimal lumen diameter

SECONDARY OUTCOMES:
device-related ischemic events | Clinical follow up at 30 days, 6, 9, 12 and 24 months after the procedure
  including cardiovascular death, target vessel related myocardial infarction and ischemia-driven revascularization
patient-related ischemic events | Clinical follow up at 30 days, 6, 9, 12 and 24 months after the operation
  all myocardial infarction , any revascularization and all-cause death
ARC（Academic Research Consortium） defined target vessel thrombus events | Clinical follow up at 30 days, 6, 9, 12 and 24 months after the operation
  definite, probable and possible target vessel thrombus

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yu, MD, Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No